CLINICAL TRIAL: NCT00935324
Title: CK18-Fragments as Tools for Evaluating Diagnosis, Biological Activity, and Prognosis of Graft-Versus-Host Disease
Brief Title: The Role of CK18F in Predicting Graft-Versus-Host Disease (GvHD)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Collaborators: University of Regensburg (Other)
Responsible Party: Prof. Dr. Peter Dreger, University of Heidelberg, Germany
Other Study IDs: HD/R-01
Record Dates: First submitted 2009-07-08; First posted 2009-07-09 (Estimated); Last update posted 2009-07-09 (Estimated); Status verified 2009-07

CONDITIONS: Allo-SCT
Keywords: allo-SCT, GvHD, CK18-F
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Group A (patients scheduled for allo-SCT): 5ml serum (~25 times), 7,5ml EDTA (~25 times) Group B (healthy volunteers): 30ml blood once
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group A: patients following allo-SCT: Patients scheduled for allo-SCT fulfilling all inclusion criteria
- Group B - healthy controls: healthy voluntary blood donors

SUMMARY:
Prospective, within-subject controlled study on multiple subject groups to evaluate the meaning of CK18-fragments in the diagnosis, biological activity and prognosis of graft-versus-host disease (GvHD). Groups consist of patients scheduled for allogenic stem cell transplantation (allo-SCT) (Group A) and healthy voluntary blood donors (Group B).

DETAILED DESCRIPTION:
Given the difficulties in assessing diagnosis, severity and biological activity of GvHD by clinical means only, objective parameters for specific GvHD assessment are highly desirable. Criteria for appropriate GvHD biomarkers have recently been defined, thereby stating that suitable validated markers for monitoring of chronic GvHD are still lacking. CK18-F is the first marker that mirrors the pathogenetic endpoint of GvHD i.e. GvHD-induced apoptotic activity in critical epithelial organs (bowel and liver). It represents a new class of GvHD markers which are complementary to the previously recognized immune activation parameters and might thereby be valuable for establishing serological signatures diagnostic for GvHD. This marker may allow distinguishing active GvHD from irreversible end organ damage and other clinical conditions commonly observed after transplant.

The aim of this study is to evaluate if diagnostic and therapeutic decisions in the clinical management of hepato-intestinal GvHD may be based on the measurement of CK18-F levels.

ELIGIBILITY:
Inclusion Criteria:

Group A:

* admission for allogenic SCT
* age >= 18 years
* ability of subject to understand character and individual consequences of this clinical trial
* written informed consent

Group B:

* healthy male of female
* age >= 18 years
* ability of subject to understand character and individual consequences of this clinical trial
* written informed consent

Exclusion Criteria:

Group A:

no specific exclusion criteria

Group B:

* prolonged bleeding, hemorrhagic diathesis or other indications for clotting disorders in the medical history
* prolonged or intense menses in females
* any other current medical condition or previous disease which in the opinion of investigator may influence subject safety or interfere with the study objective
* intake of any study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for allo-SCT
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2009-02; Primary Completion 2011-03 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
Group A: Prediction of imminent GvHD Group B: To assess the levels of serum CK18-F | Group A: after allo-SCT for 1 years or until GvHD occures

SECONDARY OUTCOMES:
Response to therapy | 3, 7 and 14 days after start of immunosuppressive therapy for hepato-intestinal GvHD
other serum markers such as sCD25, sCD40L, sFASL, sFAS, cytochrome C, sCD141 correlate with the achievement of complete responses | after allo-SCT for 1 year or until GvHD occurres
CK18-F levels in the absence of a clinically diagnosed GvHD | after allo-SCT for one year

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Luft, MD, Principal Investigator — Heidelberg University
Locations (1):
- University of Heidelberg, Heidelberg, Germany